CLINICAL TRIAL: NCT00683553
Title: A Phase I, Randomized, Double-Blind, Dose Escalation Trial of the Safety and Pharmacokinetics of a Single Intravenous Injection of I5NP in Patients at High Risk of Acute Kidney Injury Undergoing Major Cardiovascular Surgery
Brief Title: A Dose Escalation and Safety Study of I5NP to Prevent Acute Kidney Injury (AKI) in Patients at High Risk of AKI Undergoing Major Cardiovascular Surgery (QRK.004)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of an available patient population
Sponsor: Quark Pharmaceuticals (Industry)
Responsible Party: Mike Johnston, Director, Regulatory Affairs, Quark Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: QRK.004
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Acute Renal Failure; Acute Kidney Injury
Keywords: Acute Renal Failure; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I5NP drug (Experimental)
  Interventions: Drug: I5NP
- Placebo (Placebo Comparator)
  Interventions: Drug: I5NP; Drug: Placebo

INTERVENTIONS:
Drug: I5NP — Single IV injection of experimental drug given in escalated doses at 0.5, 1.5, 5.0 and 10 mg/kg doses to different patients
  Other Names: QPI-1002
Drug: Placebo — Single IV injection of saline
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, dose escalation, safety and pharmacokinetic study. The study will be conducted in approximately 10 sites in the United States. Up to 48 patients at high risk for AKI (CCF score ≥ 5 OR an estimated GFR (eGFR) <60 mL/min/1.73 m2) who have undergone major cardiovascular surgery will participate. Patients will receive a single IV injection of I5NP or placebo following cardiovascular surgery. I5NP will be administered 4 hours (+/- 30 minutes) following removal of the cardiopulmonary bypass machine (CBM).

The duration of the study is approximately 44 days, inclusive of a 14 day screening period. Patients will be contacted by phone at 6 and 12 months for follow-up questions. Patient visits are screening, day of surgery, hospital in-patient Days 1, 2, 3 - 5 and Day 7 or hospital discharge. Safety follow-up will continue until 30 days post-surgery. 2 phone calls will be made at 6 and 12 months after date of surgery.

DETAILED DESCRIPTION:
The drug (I5NP) is a small interfering RNA that is being developed to protect patients from acute kidney injury after cardiac bypass surgery. This study will test the safety of I5NP and measure how long the drug stays in the blood stream after injection. This study is not meant to test if I5NP protects kidneys from the damage that may occur in rare cases during surgery. Another purpose of this dose escalation study is to find out the right dose of the experimental drug to be given to study subjects in future studies. Even though there were no harmful effects seen in the animals tested, we do not know what side effects the experimental drug might cause in humans.

ELIGIBILITY:
Inclusion Criteria (before surgery):

* Patient age between 21 years and 85 years old
* Patient is capable of giving consent
* Patient is willing and able to comply with the visit schedule and study procedures including post-hospitalization discharge follow-up
* Patient is undergoing any major cardiac or vascular surgery requiring the use of cardiopulmonary bypass machine (CBM)
* Patient has a cumulative score of ≥ 5 on the Cleveland Clinic Foundation (CCF) Acute Kidney Injury (AKI) risk factor scale OR the patient has an estimated GFR (eGFR) <60 mL/min/1.73 m2, as determined from the simplified (4-variable) MDRD (Modification of Diet in Renal Disease) equation at the time of the Screening/Baseline examination
* The patient reports that they are up to date and have had normal findings on their age- and sex-appropriate cancer screening, per American Cancer Society guidelines, for breast cancer, cervical cancer, rectal cancer, and prostate cancer. If a patient is not up to date, the relevant screening test must be performed and a normal result documented prior to dosing.

Inclusion Criteria (during surgery):

* Patient must have been on cardiopulmonary bypass machine (CBM)

Inclusion Criteria (after surgery):

* Patient must be in the ICU for dosing to facilitate study procedures including PK blood draws and PK urine sampling

Exclusion Criteria (before surgery):

* Patient has had cancer or may be predisposed due to a family history of:

  * a clinical syndrome predisposing to malignancy, such as Familial Polyposis Coli, Von Hippel Landau disease (associated with renal cell cancers and renal cysts) and Li-Fraumeni syndrome (associated with inherited mutations of the p53 tumor-suppressor gene)
  * the same malignancy in two or more first- or second-degree relatives
* Patient has a history of any abnormality on chest X-ray that could represent a malignancy
* Patient has a clinically significantly elevated pancreatic and/or hepatic enzyme level, defined as any grade 2, 3 or 4 value according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), version 3.0
* Women of childbearing potential are to be excluded from this study. Every female subject is considered of childbearing potential unless she has had sterilization surgery, or is post-menopausal.

  * Women 21-59, post-menopausal is defined as no menses for at least 12 months and an elevated follicle stimulating hormone (FSH) level.
  * Women 60-85, post-menopausal is defined as no menses in at least 12 months.
* Patient has participated in a study of an experimental therapy in the last 30 days
* Patient is currently receiving immunosuppressive therapy [this criterion does NOT apply to topical steroids and inhalation steroids for chronic obstructive pulmonary disease (COPD) and/or asthma]
* Pre-operative extracorporeal membrane oxygenation
* Patient has Intra-Arterial Balloon Pump (IABP) or other Left Ventricular Assist Device (LVAD)
* Evidence that patient is experiencing possible AKI prior to surgery, defined as a > 1.5 times increase in serum creatinine from screening to any time prior to surgery
* Patient has comfort measures only or do not resuscitate (DNR) status
* Patient is participating in a concurrent interventional study
* Patient has received intravenous contrast material < 24 hours prior to surgery
* In the opinion of the investigator a pre-operative concomitant disease or clinical/laboratory finding that significantly raises the risk of complications in the post-operative period and therefore precludes dosing of the patient

Exclusion Criteria (during surgery):

* In the opinion of the investigator, an intra-operative complication has occurred that significantly raises the risk of complications in the post operative period and therefore precludes dosing of the patient

Exclusion Criteria (after surgery):

* In the opinion of the investigator, a complication has occurred in the post-operative period at any time prior to dosing that significantly raises the risk of further complications and therefore precludes dosing of the patient

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Number of Dose Limiting Toxicities (DLTs) observed among 4 cohorts of 6-12 patients per cohort | Reviewed at the conclusion of each cohort
Pharmacokinetics | Immediately following injection through 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Martin S. Polinsky, M.D., Study Director — Quark Pharmaceuticals
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - George Washington University, Washington D.C., District of Columbia
  - Washington University, St Louis, Missouri
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Heart Institute, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Texas, Houston, Texas
  - University of Virginia School of Medicine, Charlottesville, Virginia